CLINICAL TRIAL: NCT05074758
Title: Characterization of the microVAScular Dysfunction in COvid-19 ARDS
Acronym: VASCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210693; 2021-A01339-32 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2021-07-19; First posted 2021-10-12 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: ARDS, Human; COVID-19 Acute Respiratory Distress Syndrome
Keywords: pulmonary biological markers; alveolar dead-space; circulating endothelial cells
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples citrated tubes blood samples EDTA tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-COVID-19 ARDS patients: 20 patients with acute respiratory distress syndrome (ARDS) unrelated to COVID-19
  Interventions: Diagnostic Test: alveolar dead-space quantification; Diagnostic Test: Coagulation activation and impaired fibrinolysis explorations; Diagnostic Test: Endothelial activation / endothelial senescence
- COVID-19 ARDS patients: 20 patients with acute respiratory distress syndrome (ARDS) linked to COVID-19
  Interventions: Diagnostic Test: alveolar dead-space quantification; Diagnostic Test: Coagulation activation and impaired fibrinolysis explorations; Diagnostic Test: Endothelial activation / endothelial senescence

INTERVENTIONS:
Diagnostic Test: alveolar dead-space quantification — measurement of alveolar dead-space based on volumetric capnography
Diagnostic Test: Coagulation activation and impaired fibrinolysis explorations — blood sampling:
  * Fibrinolytic components
  * NETs components
  * Elastase-derived fragments of proteins of interest
Diagnostic Test: Endothelial activation / endothelial senescence — circulating endothelial cells, E-selectin, endoglin, LVEF-A, LVEFR-2, Angiopoietin -1 and -2, cKit and SDF-1 Willebrand factor (activity, antigen, multimeric analysis )

SUMMARY:
The primary endpoint of this research is to establish that the alveolar dead space is significantly higher in patients with COVID-19 ARDS, compared to patients with non-COVID-19 ARDS.

Secondarily, the investigators want to establish the prognostic value of the alveolar-dead space (measured iteratively) in patients with COVID-19 and non-COVID-19 ARDS, to establish the respective influences of the biological parameters of endothelial damage, of the biological parameters of coagulopathy, of the parameters set on the artificial ventilator on the value of the alveolar dead space; in ARDS patients with COVID-19 and non-COVID-19 ARDS, to establish the prognostic value of the laboratory parameters of endothelial damage and coagulopathy in patients with COVID-19 and non-COVID-19 ARDS.

DETAILED DESCRIPTION:
Endothelial damage and coagulation activation at the lung microvascular level may play an important role in the physiopathology of the COVID-19 ARDS. The project aims to prospectively investigate both bedside pulmonary physiological markers and biological markers of coagulopathy and endothelial dysfunction in COVID-19 and non-COVID-19 ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Invasive mechanical ventilation in place for less than 48 hours
* Severe or moderate ARDS (defined according to the Berlin classification)
* Virological confirmation by PCR of SARS-CoV-2 infection (ARDS COVID-19)
* Lack of virological confirmation by PCR of SARS-CoV-2 infection (ARDS not linked to COVID-19)
* Patient information

Exclusion Criteria:

* Massive pulmonary embolism
* Chronic respiratory failure under long-term oxygen therapy
* Dying patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate or severe ARDS linked or not with covid-19
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of alveolar dead space | Up to 28 days
  Recording the exhaled CO2 curve (side-stream capnography method) and volume curve, as determined by the mechanical ventilator, and computing the signals with the arterial CO2 partial pressure, reflecting the partial pressure of CO2 in the alveoli participating in gas exchanges), determined on arterial blood gas (ABG) sampling.

SECONDARY OUTCOMES:
Prognostic value of the alveolar dead space (measured iteratively) | 20 days
  To establish the link between alveolar dead-space values and Day 20 mortality
Prognostic value of the alveolar dead space (measured iteratively) | 28 days
  To establish the link between alveolar dead-space values and Day 20 mortality and Day-28 invasive ventilator-free days.
Level of circulating endothelial cells | Up to 28 days
  To describe the biological parameters of endothelial damage and prognostic value
Level of progenitor cells | Up to 28 days
  To describe the biological parameters of endothelial damage and prognostic value
Level of circulating stem cells | Up to 28 days
  To describe the biological parameters of endothelial damage and prognostic value
Level of endothelial proteomics | Up to 28 days
  To describe the biological parameters of endothelial damage and prognostic value
Level of D-dimers | Up to 28 days
  To describe the biological parameters of endothelial damage and prognostic value
Level of Willebrand Factor | Up to 28 days
  To describe the biological parameters of endothelial damage and prognostic value
Level of components of the fibrinolytic system | Up to 28 days
  To describe the biological parameters of endothelial damage and prognostic value
Level of fragments of plasminogen | Up to 28 days
  To describe the biological parameters of endothelial damage and prognostic value
Level of the components of the NETs (Neutrophil Extracellular Traps) | Up to 28 days
  To describe the biological parameters of endothelial damage and prognostic value
Survival rate | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Diehl, PhD, Study Chair — AP-HP, Hôpital Européen Georges Pompidou, Paris
Locations (1):
- Hôpital européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement. Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Diehl JL, Peron N, Chocron R, Debuc B, Guerot E, Hauw-Berlemont C, Hermann B, Augy JL, Younan R, Novara A, Langlais J, Khider L, Gendron N, Goudot G, Fagon JF, Mirault T, Smadja DM. Respiratory mechanics and gas exchanges in the early course of COVID-19 ARDS: a hypothesis-generating study. Ann Intensive Care. 2020 Jul 16;10(1):95. doi: 10.1186/s13613-020-00716-1. PMID 32676824
- [Background] Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020 Jul 9;383(2):120-128. doi: 10.1056/NEJMoa2015432. Epub 2020 May 21. PMID 32437596